CLINICAL TRIAL: NCT04582695
Title: Integrated Early Intervention for Alcohol Use Disorder and Posttraumatic Stress Disorder Following Sexual Assault
Brief Title: Early Intervention Following Sexual Assault
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00099114; 1K23AA028055 (NIH)
Record Dates: First submitted 2020-09-28; First posted 2020-10-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ptsd; Alcohol Use Disorder; Sexual Assault and Rape
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Cognitive Behavioral Therapy; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Exposure Therapy (Active Comparator)
  Interventions: Behavioral: Written Exposure Therapy
- Written Exposure Therapy Integrated with Cognitive Behavioral Therapy for Alcohol Use Disorder (Experimental)
  Interventions: Behavioral: Written Exposure Therapy Integrated with Cognitive Behavioral Therapy for Alcohol Use Disorder

INTERVENTIONS:
Behavioral: Written Exposure Therapy Integrated with Cognitive Behavioral Therapy for Alcohol Use Disorder — Participants will receive 5 to 6 weeks of an integrated behavioral therapy that address posttraumatic stress disorder and alcohol use disorder. Sessions will be 60 minutes in length. It will include written exposure therapy, which involves writing about their experience of sexual assault for 30 minutes. In addition, they will receive 20 minutes of intervention focused on cognitive behavioral therapy for alcohol use disorder which involves learning skills to cope with alcohol cravings and behavior (e.g., challenging thoughts, problem solving).
  Arms: Written Exposure Therapy Integrated with Cognitive Behavioral Therapy for Alcohol Use Disorder
Behavioral: Written Exposure Therapy — Participants will receive 5 to 6 weeks of written exposure therapy, which involves writing about their experience of sexual assault for 30 minutes.
  Arms: Written Exposure Therapy

SUMMARY:
This study is for women who have experienced a sexual assault in the past six weeks and use alcohol. The research involves completing a five week behavioral treatment for stress and alcohol use. Participants will complete surveys during visits. Participants may also be asked to complete brief daily assessments on their smart phones.

DETAILED DESCRIPTION:
The primary objective of the proposed Stage IA/IB study is to establish feasibility of an integrated cognitive-behavioral intervention for reducing alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD) symptoms among women who experienced a sexual assault within the past six weeks. The intervention will be tested in an open label trial to make final modifications to evaluate feasibility, acceptability, and preliminary efficacy of the five to six week integrated intervention with standardized repeated measures during a one-month follow-up. Next, a pilot randomized controlled trial will be conducted among 54 recent sexual assault victims to evaluate feasibility and preliminary efficacy in reducing AUD severity and PTSD symptoms. Ecological momentary assessments (EMA) will be used to assess alcohol use, craving, and affect during the five-week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Female; any race or ethnicity; age 18 to 65 years old.
* Sexual assault that occurred within the past 12 months.
* Subjects must be able to comprehend English.
* A score of 3 or greater on the Alcohol Use Disorders Identification Test (AUDIT-C) screen.
* A score of 31 or greater on the Posttraumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders (PCL-5). Subjects may also meet criteria for an alcohol use disorder, previous history of posttraumatic stress disorder, mood disorder (except bipolar affective disorder, see Exclusion Criteria) or other anxiety disorders (panic disorder, agoraphobia, social phobia, generalized anxiety disorder, or obsessive-compulsive disorder). The inclusion of subjects with affective and other anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with AUD and PTSD (Norman et al., 2018; Zinzow et al., 2012). Subjects may meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for another substance use disorder if AUD is the primary substance of choice.
* Must consent to complete all treatment and follow-up visits.

Exclusion Criteria:

* Lack of any memory of the sexual assault
* Subjects meeting the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for a history of or current psychotic, bipolar, dissociative identify disorder, or a current eating disorder, as the study protocol may be therapeutically insufficient.
* Subjects experiencing significant withdrawal symptoms, as evidence by a score of 10 or more on the Clinical Institute Withdrawal Assessment of Alcohol (CIWA). These subjects will be referred for clinical detoxification and may be re-assessed for study eligibility after medically supervised detoxification has been completed.
* Individuals considered an immediate suicide risk, with current suicidal ideation and intent.
* Individuals who attempted suicide in the past month. These individuals will be referred directly for treatment.
* Individuals on psychotropic medications must be stabilized on it for at least two weeks prior to beginning the study.
* Any other medical or psychiatric conditions that the investigators believe may compromise the individual's ability to safely participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women only
Enrollment: 60 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Percent Drinking Days on The Time Line Follow-Back | Participants will report on drinking during the 30 days prior to initiation of the study, and every day until study completion completion of study visits, approximately six weeks.
  The Time Line Follow Back (TLFB) will be used to assess heavy drinking in the past 30-days. This calendar-assisted interview yielded estimates in terms of the number of standard drinks consumed daily in the past 30 days used to obtain retrospective self-report of alcohol use by using a calendar and other memory prompts to stimulate recall.
Change in number of standard drinks per drinking day on The Time Line Follow-Back | Participants will report on drinking during the 30 days prior to initiation of the study, and ever day until completion of study visits, approximately six weeks.
  The Time Line Follow Back (TLFB) will be used to assess heavy drinking in the past 30-days and use. This calendar-assisted interview yielded estimates in terms of the number of standard drinks consumed daily in the past 30 days used to obtain retrospective self-report of alcohol use by using a calendar and other memory prompts to stimulate recall.
Change in Posttraumatic Stress Disorder Symptoms on The Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders (PCL-5) | Baseline and after completion of study visits, approximately six weeks.
  Participants will be asked to complete the 20-item Posttraumatic Checklist for Diagnostic and Statistical Manual of Mental Disorders (PCL-5) to measure traumatic stress symptoms corresponding with the Diagnostic and Statistical Manual of Mental Disorders -5 PTSD criteria. Items are rated on a five-point Likert scale ranging from 0 (Not at all) to 4 (Extremely) with higher scores indicating greater traumatic stress symptoms. Total scores will be used.
Change in Posttraumatic Stress Disorder Symptoms on The Clinician-Administered Posttraumatic Stress Disorder Scale for the Diagnostic and Statistical Manual of Mental Disorders | Baseline and after completion of study visits, approximately six weeks.
  The Clinician-Administered Posttraumatic Stress Disorder Scale for the Diagnostic and Statistical Manual of Mental Disorders (CAPS-5) is the gold standard in Posttraumatic Stress Disorder (PTSD) assessment. It is a structured 30-minute interview that can be used to diagnosis PTSD. Items focus on symptom presence, onset and duration of symptoms, subjective distress, impact on functioning, and symptom improvement.

SECONDARY OUTCOMES:
Change in Depression Symptoms on The Patient Health Questionnaire-9. | Baseline and after completion of study visits, approximately six weeks.
  The Patient Health Questionnaire-9 is a widely used self-report measure for attitudes and symptoms of depression. The PHQ-9 includes 9 self-report items. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 27. A total score of 0-4 is considered minimal range, 5-9 is mild, 10-14 is moderate, 15-19 is moderately severe, and 20 or more is severe.
Change in Anxiety Symptoms on The Beck Anxiety Inventory | Baseline and after completion of study visits, approximately six weeks.
  The Beck Anxiety Inventory (BAI) assesses symptoms of anxiety via 21-item self-report. The BAI reliability discriminates anxiety-disordered from non-anxiety disordered patients and demonstrates excellent convergence with related anxiety scales. The values for each item are summed yielding an overall or total score for all 21 symptoms that can range between 0 and 63 points. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and; 26 - 63 as "Severe".
Change in Percent Days Using Substances on The Time Line Follow-Back | Participants will report on substance use during the 30 days prior to initiation of the study, and every day until study completion completion of study visits, approximately six weeks.
  The Time Line Follow-Back will be used to assess illicit substance use in the past 30-days. This calendar-assisted interview yielded estimates in terms of self-report of substance use by using a calendar and other memory prompts to stimulate recall.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783

DOCUMENTS (1):
  • Informed Consent Form (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT04582695/ICF_000.pdf